CLINICAL TRIAL: NCT00909103
Title: Computer-aided Diagnosis of Endoscopic Ultrasound Elastography Used in the Differentiation of Focal Pancreatic Masses
Brief Title: Endoscopic Ultrasound Elastography in Pancreatic Masses
Acronym: EUS-EG
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Odense University Hospital (Other); Institut Paoli-Calmettes (Other); San Raffaele University Hospital, Italy (Other); UCL (Univ), Brussels, Belgium (Unknown); Glasgow Royal Infirmary (Other); Caritas-Krankenhaus Bad Mergentheim (Other); University of Bergen (Other); University of Witten/Herdecke (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Adrian Saftoiu, University of Medicine and Pharmacy Craiova, Romania
Other Study IDs: EUS-EG001; EUS-EG-UMFCV-RO
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Pancreatic Adenocarcinoma; Chronic Pancreatitis
Keywords: Endoscopic Ultrasound Elastography; Pancreatic adenocarcinoma; Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pathology samples obtained from duodeno-pancreatectomies or caudal pancreatectomies done with curative intent, as well as microhistological fragments obtained through EUS-FNA biopsy processed by paraffin embedding
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pancreatic adenocarcinoma: Patients diagnosed with solid pancreatic adenocarcinoma masses, with cytological / histological confirmation
- Chronic pancreatitis: Patients diagnosed with solid pancreatic tumor masses with all the criteria fulfilled to exclude pancreatic cancer

SUMMARY:
The aim of the study is to assess elastography during EUS examinations of focal pancreatic masses, and to consequently differentiate benign versus malignant pancreatic masses in a prospective multi-center design.

DETAILED DESCRIPTION:
Ultrasound elastography is a recent ultrasound method used for the calculation of tissue elasticity distribution in real-time. The method allows the reconstruction of tissue elasticity (i.e. the elasticity modulus) and reveals directly the physical properties of the tissue, consequently showing different tissue hardness patterns that are determined by diseases. Tissue elastography can be easily performed real-time with conventional probes, including the linear EUS probes used for the examination of the pancreas. The calculation of tissue elasticity distribution is performed in real-time and the examination results are represented as transparent overlay colour images overimposed on the conventional gray-scale B-mode images.

Ultrasound elastography was previously used for the diagnosis of breast lesions, prostate cancer and thyroid nodules. However, the value of endoscopic ultrasound elastography for the diagnosis of pancreatic focal masses is not clear for the current moment, as some authors couldn't differentiate benign and malignant pancreatic tumors. Moreover, the intense fibrotic reaction and calcifications in chronic pancreatitis induce strain differences, and it is not clear if elastography is sensitive enough to detect them.

The study protocol is based on a semi-quantitative approach of EUS elastography data (movies) consisting of characterization of manually user-defined regions of interest, based on the hue histograms of the individual focal masses. Due to the inherent bias induced by selection of images from a dynamic sequence of EUS elastography, we have previously reported on the utility of using computer-aided diagnosis by averaging images from a dynamic sequence of EUS elastography. A special plugin (based on the ImageJ software, NIH, Bethesda, MD, USA) is used to compute hue histograms on average EUS elastography images, while the hue histograms values for each patient (0 to 255 values) are further used to classify the patients with benign and malignant lesions.

Ultrasound elastography will be performed during an usual EUS examination (7.5 MHz frequency), with two movies of 10 seconds recorded on the embedded HDD in order to minimize variability and to increase repeatability of acquisition. A two panel image with the usual conventional gray-scale B-mode EUS image on the right side and with the elastography image on the left side will be used. The region of interest will be preferably larger than the focal mass, in order to include the surrounding structures. In order to minimize the human bias, all the post-processing and computer analysis of digital movies will be performed within the IT Center in Craiova, with all programmers and statisticians being blinded to the clinical, pathological and imaging data, with the exception of the average hue histogram values calculated from a second region of interest manually traced around the focal mass.

The study design is prospective, blinded and multi-center, comparing endoscopic ultrasound elastography (EUS-EG) results for the detection and characterization of focal pancreatic masses by using artificial intelligence techniques, in comparison with the gold standard represented by pathology. The study will be performed with the approval of the institutional board review of each center.

ELIGIBILITY:
Inclusion criteria

* Patients diagnosed with solid pancreatic tumor masses, with cytological / histological confirmation
* Age 18 to 80 years old, men or women
* Signed informed consent for EUS with elastography and FNA biopsy

Exclusion criteria

* Prior surgical treatment with curative intent or chemo-radiotherapy
* Patients diagnosed with mucin producing tumors, pancreatic cystic tumors, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The diagnosis of chronic pancreatitis will be based on the clinical information (history of alcohol abuse, previous diagnosis of chronic pancreatitis or diabetes mellitus), as well as a combination of imaging methods (ultrasound, CT and EUS). At least four criteria of chronic pancreatitis during EUS will be considered for the positive diagnosis.
  A positive cytological diagnosis will be taken as a final proof of malignancy of the pancreas mass. The diagnoses obtained by EUS-FNA will be further verified either by surgery or during a clinical follow-up of at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Value of endoscopic ultrasound elastography for the differential diagnoses of pancreatic masses. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Saftoiu, Professor, Study Director — University of Medicine and Pharmacy Craiova, Romania
Locations (18):
- Belgium (2):
  - Erasme University, Brussels
  - Universite Chatolique Louvain, Brussels
- Denmark (2):
  - Gentofte University Hospital, Copenhagen
  - University Hospital, Odense
- Institute Paoli Calmettes, Marseille, France
- Germany (6):
  - Caritas-Krankenhaus, Bad Mergentheim
  - St. Josef Hospital, Bochum
  - SRH Klinik, Gera
  - University Clinic Mainz, Mainz
  - Dr.Horst-Schmidt-Klinik, Wiesbaden
  - HELIOS Klinikum Wuppertal, University of Witten/Herdecke, Wuppertal
- Hospital San Raffaele, Milan, Italy
- Erasme Medisch Centrum, Rotterdam, Netherlands
- University of Haukeland, Bergen, Norway
- University of Medicine and Pharmacy Craiova, Craiova, Romania
- University Hospital Santiago, Santiago, Spain
- United Kingdom (2):
  - Glasgow Royal Infirmary, Glasgow
  - Newcastle Upon Tyne Hospitals, Newcastle

REFERENCES:
- [Background] Frey H. [Realtime elastography. A new ultrasound procedure for the reconstruction of tissue elasticity]. Radiologe. 2003 Oct;43(10):850-5. doi: 10.1007/s00117-003-0943-2. German. PMID 14605701
- [Background] Ophir J, Alam SK, Garra B, Kallel F, Konofagou E, Krouskop T, Varghese T. Elastography: ultrasonic estimation and imaging of the elastic properties of tissues. Proc Inst Mech Eng H. 1999;213(3):203-33. doi: 10.1243/0954411991534933. PMID 10420776
- [Background] Itoh A, Ueno E, Tohno E, Kamma H, Takahashi H, Shiina T, Yamakawa M, Matsumura T. Breast disease: clinical application of US elastography for diagnosis. Radiology. 2006 May;239(2):341-50. doi: 10.1148/radiol.2391041676. Epub 2006 Feb 16. PMID 16484352
- [Background] Miyanaga N, Akaza H, Yamakawa M, Oikawa T, Sekido N, Hinotsu S, Kawai K, Shimazui T, Shiina T. Tissue elasticity imaging for diagnosis of prostate cancer: a preliminary report. Int J Urol. 2006 Dec;13(12):1514-8. doi: 10.1111/j.1442-2042.2006.01612.x. PMID 17118027
- [Background] Rago T, Santini F, Scutari M, Pinchera A, Vitti P. Elastography: new developments in ultrasound for predicting malignancy in thyroid nodules. J Clin Endocrinol Metab. 2007 Aug;92(8):2917-22. doi: 10.1210/jc.2007-0641. Epub 2007 May 29. PMID 17535993
- [Background] Janssen J, Schlorer E, Greiner L. EUS elastography of the pancreas: feasibility and pattern description of the normal pancreas, chronic pancreatitis, and focal pancreatic lesions. Gastrointest Endosc. 2007 Jun;65(7):971-8. doi: 10.1016/j.gie.2006.12.057. PMID 17531630
- [Background] Saftoiu A, Vilmann P, Ciurea T, Popescu GL, Iordache A, Hassan H, Gorunescu F, Iordache S. Dynamic analysis of EUS used for the differentiation of benign and malignant lymph nodes. Gastrointest Endosc. 2007 Aug;66(2):291-300. doi: 10.1016/j.gie.2006.12.039. PMID 17643702
- [Derived] Saftoiu A, Vilmann P, Gorunescu F, Janssen J, Hocke M, Larsen M, Iglesias-Garcia J, Arcidiacono P, Will U, Giovannini M, Dietrich CF, Havre R, Gheorghe C, McKay C, Gheonea DI, Ciurea T; European EUS Elastography Multicentric Study Group. Efficacy of an artificial neural network-based approach to endoscopic ultrasound elastography in diagnosis of focal pancreatic masses. Clin Gastroenterol Hepatol. 2012 Jan;10(1):84-90.e1. doi: 10.1016/j.cgh.2011.09.014. Epub 2011 Oct 1. PMID 21963957
- [Derived] Saftoiu A, Vilmann P, Gorunescu F, Janssen J, Hocke M, Larsen M, Iglesias-Garcia J, Arcidiacono P, Will U, Giovannini M, Dietrich C, Havre R, Gheorghe C, McKay C, Gheonea DI, Ciurea T; European EUS Elastography Multicentric Study Group. Accuracy of endoscopic ultrasound elastography used for differential diagnosis of focal pancreatic masses: a multicenter study. Endoscopy. 2011 Jul;43(7):596-603. doi: 10.1055/s-0030-1256314. Epub 2011 Mar 24. PMID 21437851
- See also: Related Info — http://elastostudy.umfcv.ro/